

## CONSENT TO PARTICIPATE IN RESEARCH

Bibliotherapy for Improving Caregiving Appraisal among Informal Caregivers of People with Dementia: A Pilot Randomized Controlled Trial

| Reference Number: HSEARS20181120001 |
|---|
| I hereby consent to participate in the captioned research conducted by Dr. Daphne Cheung. |
| I understand that information obtained from this research may be used in future research and published. However, my right to privacy will be retained, i.e. my personal details will not be revealed. |
| The procedure as set out in the attached information sheet has been fully explained. I understand the benefit and risks involved. My participation in the project is voluntary. |
| I acknowledge that I have the right to question any part of the procedure and can withdraw at any time without penalty of any kind. |
| Name of participant |
| Signature of participant |
| Name of Parent or Guardian (if applicable) |
| Signature of Parent or Guardian (if applicable) |
| Name of researcher Dr. Daphne Cheung |
| Signature of researcher |
| Date |

## **INFORMATION SHEET**

## Bibliotherapy for Improving Caregiving Appraisal among Informal Caregivers of People with Dementia: A Pilot Randomized Controlled Trial

You are invited to participate in a study conducted by Dr. Daphne Cheung, who is a research assistant professor of School of Nursing in The Hong Kong Polytechnic University. The project has been approved by the Human Subjects Ethics Sub-committee (HSESC) of The Hong Kong Polytechnic University (HSESC Reference Number: HSEARS20181120001).

The aim of this study is to explore the feasibility of the intervention protocol, and the efficacy of bibliotherapy on improving caregiving appraisal, coping, positive aspects of caregiving and psychological well-being for informal caregivers of people with dementia in China. The study will involve completing a questionnaire before group allocation, which will take you about half an hour. After completing the questionnaire, you will either be allocated to the intervention group or control group randomly. For participants in the intervention group, they will receive bibliotherapy without withdrawing from the usual care. They will be asked to read the designated manual (consists of nine chapters) within a recommended period of time (over 9 weeks). Weekly telephone follow-up will also be given to them. They will be asked not to share the reading materials with others before the completion of the intervention. For participants in the control group, they will only receive usual care provided by the community health professionals. They will also be asked not to communicate with participants in the intervention group during the intervention period. After the completion of the intervention, participants in both groups will be asked to fill in the same set of questionnaires as pre-intervention.

The testing should not result in any undue discomfort. All information related to you will remain confidential and will be identifiable by codes only known to the researcher.

You have every right to withdraw from the study before or during the measurement without penalty of any kind.

If you would like to obtain more information about this study, please contact Dr Daphne Cheung (tel. no.: +852 97172170 / email: daphne.cheung@polyu.edu.hk).

If you have any complaints about the conduct of this research study, please do not hesitate to contact Miss Cherrie Mok, Secretary of the Human Subjects Ethics Sub-Committee of The Hong Kong Polytechnic University in writing (c/o Research Office of the University) stating clearly the responsible person and department of this study as well as the HSESC Reference Number.

Thank you for your interest in participating in this study.

Dr Daphne Cheung Principal Investigator

> Hung Hom Kowloon Hong Kong 香港 九龍 紅磡 Tel 電話 (852) 2766 5111 Fax 傳真 (852) 2784 3374 Email 電郵 polyu@polyu.edu.hk Website 網址 www.polyu.edu.hk